CLINICAL TRIAL: NCT06559423
Title: Combined Non-ablative Er:YAG Laser and High Intensity Tesla Magnetic Stimulation (HITS) for Treatment of Female Urinary Incontinence: A Single-centre, Single-arm Pilot Study
Brief Title: Combined Non-ablative Er:YAG Laser and Magnetic Stimulation for Treatment of Female Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zdravstveni Zavod Štrumbelj (Other)
Collaborators: Fotona d.o.o. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Study Laser + HITS
Record Dates: First submitted 2024-08-09; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Stress Urinary Incontinence; Urinary Incontinence
Keywords: stress urinary incontinence; urinary incontinence; non-ablative erbium laser; magnetic stimulation; High Intensity Tesla magnetic Stimulation (HITS); combined therapy; Er:YAG laser
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser + HITS (Experimental): The treatment involved three consecutive Er:YAG laser sessions (TimeWalker® Intima Laser™, Fotona) followed by six HITS treatments (StarFormer® IntimaWave®, Fotona).
  The laser sessions were spaced one month apart, following the IncontiLase® protocol using the G-Runner robotic handpiece. The protocol included three steps: (i) intravaginal laser treatment of the anterior vaginal wall, (ii) treatment of the entire vaginal canal, and (iii) treatment of the vestibule and introitus. Each session lasted 20 minutes.
  Six weeks after the final laser treatment, patients received six HITS treatments, with two sessions per week. The HITS protocol involved increasing stimulation frequencies, each for 10 minutes, with the total session lasting 30 minutes.
  Interventions: Device: non-ablative Er:YAG laser and high intensity Tesla magnetic stimulation (HITS)

INTERVENTIONS:
Device: non-ablative Er:YAG laser and high intensity Tesla magnetic stimulation (HITS) — Patients will initially undergo three monthly intravaginal treatments with the Er:YAG laser. Six weeks after the final laser treatment, patients will receive six sessions of magnetic stimulation. During these sessions, patients will sit on a specialized chair that generates a therapeutic magnetic field.

SUMMARY:
This single-arm pilot study aims to investigate the efficacy and safety of a combined non-ablative Erbium:Yttrium-Aluminium-Garnet (Er:YAG) laser and High Intensity Tesla magnetic Stimulation (HITS) treatment for female urinary incontinence. The study involves 25 women diagnosed with mild to moderate stress or mixed urinary incontinence. Participants will receive three vaginal Er:YAG laser treatments and six HITS sessions. The primary objective is to improve symptoms of urinary incontinence, as measured by changes in scores on two questionnaires compared to baseline. Secondary objectives include improvement in sexual function, durability of improvement in urinary incontinence symptoms at 3- and 6- month follow-up, patient-reported improvement, and discomfort during treatment.

DETAILED DESCRIPTION:
The aim of this single-centre, single-arm pilot study is to investigate the combined effects of vaginal Er:YAG laser and HITS treatment on urinary incontinence (UI) in women. The study will involve 25 women suffering from mild to moderate stress urinary incontinence or mixed urinary incontinence. The aim of the study is to investigate whether the combination of non-ablative Er:YAG laser therapy and HITS can have a synergistic effect in relieving UI symptoms. Participants will undergo three sessions of intravaginal laser treatment according to the IncontiLase® Er:YAG laser protocol and six HITS sessions. The laser treatments will take place one month apart, while the HITS sessions will take place twice a week for three weeks after the last laser treatment.

Primary endpoints include improvement in UI symptoms as measured by changes in International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) and Questionnaire for Urinary Incontinence Diagnosis (QUID) scores from baseline to post-treatment. Secondary endpoints include improvement in sexual function as measured by the Female Sexual Function Index (FSFI), durability of improvement in UI symptoms 3 and 6 months after treatment, patient-reported global impression of improvement (Patient Global Impression of Improvement, PGI-I), and treatment-related discomfort as measured by the Visual Analog Scale (VAS) for pain.

The study also includes rigorous safety assessments and monitoring of adverse events or complaints during and after the treatments. Recruitment of participants will ensure that they meet certain inclusion criteria, such as adult women with a clinical diagnosis of stress or mixed UI, as well as exclusion criteria to minimize risks and improve compliance.

Statistical analysis will be performed using various tests to check the data for normality and distribution. The results of the study should provide valuable insight into the efficacy and safety of combining laser and HITS treatments for female urinary incontinence and potentially provide a new non-invasive treatment option for this condition.

ELIGIBILITY:
Inclusion Criteria:

* Adult female, 18 years of age or older
* Clinical diagnosis of stress or mixed urinary incontinence, with stress incontinence as the predominant symptom

Exclusion Criteria:

* Very severe urinary incontinence (ICIQ-UI SF score at baseline >18)
* Pregnancy
* BMI>35
* Not willing to abstain from vaginal intercourse for one week following the laser-therapy
* Acute urinary tract infections (UTIs)
* History of a genital fistula, a thin recto-vaginal septum as determined by the investigator or history of a fourth-degree laceration during screening physical exam (e.g., perineal body)
* Active sexually transmitted disease upon vaginal exam (as determined by the investigator) that precludes treatment or any other vaginal infection
* Prolapse grade 2 or higher
* History of radiotherapy for cervical or uterine cancer
* Medical condition that may interfere with participants' compliance to the protocol
* Medical condition for which the HITS and laser therapy are contraindicated
* Previous laser or HITS treatment for UI

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Efficacy of the combined laser and HITS treatment | up to 6 months after treatment
  Improvement of symptoms of stress and/or mixed urinary incontinence as measured by change in ICIQ-UI SF and QUID scores from the baseline.
Safety of the combined laser and HITS treatment | up to 6 months after treatment
  Incidence and severity of treatment-related Adverse Events

SECONDARY OUTCOMES:
Improvement of sexual function | up to 6 months after treatment
  Improvement of sexual function as measured by FSFI scores change from baseline
Durability of the effect | up to 6 months after treatment
  Improvement of the urinary incontinence symptoms measured at 3 and 6 months follow-up
Patient reported assessment of improvement | up to 6 months after treatment
  Assessed by PGI-I questionnaire
Patient reported assessment of discomfort during treatment | up to 24 hours after each laser and HITS session
  Measured by visual analog scale pain score

CONTACTS AND LOCATIONS:
Overall Officials: Tadeja Štrumbelj, MD, Principal Investigator — Zdravstveni Zavod Štrumbelj
Locations (1):
- Zdravstveni Zavod Štrumbelj, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No